CLINICAL TRIAL: NCT01863732
Title: An Extension Study to Evaluate the Sustainability of Clinical Benefits, Safety and Tolerability of Secukinumab in Patients With Active Ankylosing Spondylitis
Brief Title: Extension in AS: Sustainability of Benefits, Safety and Tolerability
Acronym: MEASURE 1 ext
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457F2305E1; 2013-001089-40 (EudraCT Number)
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-06

CONDITIONS: Spondylitis, Ankylosing
Keywords: AIN457, ankylosing spondylitis, chronic inflammatory disease, inflammatory back pain, PFS, pre-filled syringe, secukinumab, self-injection
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Secukinumab (AIN457) 75mg Grp1 (Experimental): Group 1: AIN457 75 mg plus placebo 150 mg dosed every four weeks Week 104E1 through Week 152. Starting on Week 156 (after unblinding), only AIN457 75 mg was dosed. Secukinumab in PFS for s.c. self-administration Q4W
  Interventions: Biological: Secukinumab; Other: Placebo (Pbo)
- Secukinumab (AIN457) 75 to 150mg Grp1 (Experimental): Group 1: AIN457 75 mg plus placebo 150 mg dosed every four weeks Week 104E1 through Week 152. Starting on Week 156 (after unblinding), was up titrated to AIN457 150 mg only. Secukinumab in PFS for s.c. self-administration Q4W
  Interventions: Biological: Secukinumab; Other: Placebo (Pbo)
- Secukinumab (AIN457) 150mg Grp2 (Experimental): Group 2: AIN457 150 mg plus placebo 75 mg dosed every four weeks Week 104E1 through Week 152. Starting on Week 156 (after unblinding), only AIN457 150 mg was dosed. Secukinumab in PFS for s.c. self-administration Q4W
  Interventions: Biological: Secukinumab; Other: Placebo (Pbo)
- Pbo in Core then AIN457 75mg Grp1 (Experimental): Participants were on Placebo (Pbo) in Core and then in extension randomized to Group 1: secukinumab (AIN457) 75 mg plus placebo 150 mg dosed every four weeks Week 104E1 through Week 152. Starting on Week 156 (after unblinding), only AIN457 75 mg was dosed.Secukinumab in PFS for s.c. self-administration Q4W
  Interventions: Biological: Secukinumab; Other: Placebo (Pbo)
- Pbo in Core then AIN457 75 to 150mg Grp1 (Experimental): Participants were on Placebo in Core and then in extension randomized to Group 1: secukinumab (AIN457) 75 mg plus placebo 150 mg dosed every four weeks Week 104E1 through Week 152. Starting on Week 156 (after unblinding), was up titrated to AIN457 150 mg only. Secukinumab in PFS for s.c. self-administration Q4W
  Interventions: Biological: Secukinumab; Other: Placebo (Pbo)
- Pbo in Core then AIN457 150mg Grp2 (Experimental): Participants were on Placebo (Pbo) in Core and then in extension randomized to Group 2: AIN457 150 mg plus placebo 75 mg dosed every four weeks Week 104E1 through Week 152. Starting on Week 156 (after unblinding), only AIN457 150 mg was dosed. Secukinumab in PFS for s.c. self-administration Q4W
  Interventions: Biological: Secukinumab; Other: Placebo (Pbo)

INTERVENTIONS:
Biological: Secukinumab — Group 1: secukinumab 75 mg plus placebo 150 mg or Group 2 secukinumab 150 mg plus placebo 75m dosed every four weeks Week 104E1 through Week 152. Starting on Week 156 (after unblinding), only secukinumab 75 mg or 150 mg were dosed. Secukinumab in PFS for s.c. self-administration Q4W
  Other Names: AIN457
Other: Placebo (Pbo) — Group 1: secukinumab 75 mg plus placebo 150 mg or Group 2 secukinumab 150 mg plus placebo 75m dosed every four weeks Week 104E1 through Week 152. Starting on Week 156 (after unblinding), only secukinumab 75 mg or 150 mg were dosed. Secukinumab in PFS for s.c. self-administration Q4W

SUMMARY:
This 3-year extension study aims at making available the treatment with secukinumab in prefilled syringes (PFS) to patients with ankylosing spondylitis who took part in phase III study CAIN457F2305, defined as "core study", as well as to generate additional data on the sustainability of clinical benefits, safety and tolerability during long-term administration of secukinumab.

ELIGIBILITY:
Inclusion Criteria: patients having completed the "core study" CAIN457F2305, indication for treatment extension. -- Exclusion Criteria: history of hypersensitivity to secukinumab or to any drug of similar chemical classes, use of any investigational drug other than secukinumab during the "core study" CAIN457F2305.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2013-11-06 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (53):
- United States (5):
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Jackson, Tennessee
  - Novartis Investigative Site, Kingsport, Tennessee
  - Novartis Investigative Site, Spokane, Washington
- Belgium (4):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Bulgaria (3):
  - Novartis Investigative Site, Burgas
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
- Canada (2):
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
- France (3):
  - Novartis Investigative Site, Limoges, Haute Vienne
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Paris
- Germany (7):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Nuremberg
- Italy (5):
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Torino, TO
- Mexico (4):
  - Novartis Investigative Site, Mexicali, Estado de Baja California
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Culiacán, Sinaloa
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Utrecht
- Peru (5):
  - Novartis Investigative Site, Jesus Maria, Lima region
  - Novartis Investigative Site, La Victoria, Lima region
  - Novartis Investigative Site, Pueblo Libre, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, Surquillo, Lima region
- Russia (5):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Tula
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Taiwan (2):
  - Novartis Investigative Site, Taichung, Taiwan ROC
  - Novartis Investigative Site, Kaohsiung City
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Gaziantep
  - Novartis Investigative Site, Izmir
- United Kingdom (4):
  - Novartis Investigative Site, London, England
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Baraliakos X, Van den Bosch F, Machado PM, Gensler LS, Marzo-Ortega H, Sherif B, Quebe-Fehling E, Porter B, Gaillez C, Deodhar A. Achievement of Remission Endpoints with Secukinumab Over 3 Years in Active Ankylosing Spondylitis: Pooled Analysis of Two Phase 3 Studies. Rheumatol Ther. 2021 Mar;8(1):273-288. doi: 10.1007/s40744-020-00269-6. Epub 2020 Dec 22. PMID 33351179
- [Derived] Tseng JC, Wei JC, Deodhar A, Martin R, Porter B, McCreddin S, Talloczy Z. Secukinumab Demonstrates Sustained Efficacy and Safety in a Taiwanese Subpopulation With Active Ankylosing Spondylitis: Four-Year Results From a Phase 3 Study, MEASURE 1. Front Immunol. 2020 Nov 26;11:561748. doi: 10.3389/fimmu.2020.561748. eCollection 2020. PMID 33324394
- [Derived] Kvien TK, Conaghan PG, Gossec L, Strand V, Ostergaard M, Poddubnyy D, Williams N, Porter B, Shete A, Gilloteau I, Deodhar A. Secukinumab and Sustained Reduction in Fatigue in Patients With Ankylosing Spondylitis: Long-Term Results of Two Phase III Randomized Controlled Trials. Arthritis Care Res (Hoboken). 2022 May;74(5):759-767. doi: 10.1002/acr.24517. Epub 2022 Mar 10. PMID 33227175
- [Derived] Baraliakos X, Braun J, Deodhar A, Poddubnyy D, Kivitz A, Tahir H, Van den Bosch F, Delicha EM, Talloczy Z, Fierlinger A. Long-term efficacy and safety of secukinumab 150 mg in ankylosing spondylitis: 5-year results from the phase III MEASURE 1 extension study. RMD Open. 2019 Sep 3;5(2):e001005. doi: 10.1136/rmdopen-2019-001005. eCollection 2019. PMID 31565244
- [Derived] Braun J, Baraliakos X, Deodhar A, Poddubnyy D, Emery P, Delicha EM, Talloczy Z, Porter B. Secukinumab shows sustained efficacy and low structural progression in ankylosing spondylitis: 4-year results from the MEASURE 1 study. Rheumatology (Oxford). 2019 May 1;58(5):859-868. doi: 10.1093/rheumatology/key375. PMID 30590813
- See also: Introduction to clinical research conducted by Novartis and to the results of completed studies. For the sake of transparency, objective scientific information is made publicly available in a standardised format. — http://www.novartisclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: CAIN457F2305 core study consisted of a screening period of 4 Wks before randomization followed by a treatment period of 2 years (Wk 0 through Wk 104). At Wk 104, patients continued into the extension on the same dose of AIN457. If they were on Placebo in the core then randomized to either Group 1 or 2.
Pre-assignment Details: Group 1: AIN457 75mg plus placebo 150mg dosed every 4 weeks from Wk 104E1 to Wk 152. At Wk 156 (after unblinding), only AIN457 75mg was dosed or up titrated to AIN457 150mg. Group 2: AIN457 150mg plus placebo 75mg dosed every 4 weeks from Wk 104E1 through Wk 152. At Wk 156 (after unblinding), only secukinumab 150 mg was dosed.
Groups:
- Secukinumab (AIN457) 75mg Group 1: AIN457 75 mg plus placebo to AIN457 150 mg dosed every four weeks Week 104E1 through Week 152. Starting on Week 156 (after unblinding), AIN457 75 mg was dosed or uptitration to AIN457 150 mg. Secukinumab in PFS for s.c. self-administration Q4W. Participants that up-titrated to AIN457 150 mg were counted only at the originally randomized AIN457 75 mg treatment group.
- Secukinumab (AIN457) 150mg Group 2: AIN457 150 mg plus placebo to AIN457 75 mg dosed every four weeks Week 104E1 through Week 152. Starting on Week 156 (after unblinding), only AIN457 150 mg was dosed. Secukinumab in PFS for s.c. self-administration Q4W.
- Pbo in Core Then AIN457 75mg Group 1: Participants were randomized on Placebo (Pbo) in Core and then re-randomized to Group 1: secukinumab (AIN457) 75 mg plus placebo to AIN457 150 mg dosed every four weeks Week 104E1 through Week 152. Starting on Week 156 (after unblinding), AIN457 75 mg was dosed or uptitration to AIN457 150mg. Secukinumab in PFS for s.c. self-administration Q4W. Participants that up-titrated to AIN457 150 mg were counted only at the originally randomized AIN457 75 mg treatment group.
- Pbo in Core Then AIN457 150mg Group 2: Participants were randomized on Placebo (Pbo) in Core and then re-randomized to Group 2: AIN457 150 mg plus placebo to AIN457 75 mg dosed every four weeks Week 104E1 through Week 152. Starting on Week 156 (after unblinding), only AIN457 150 mg was dosed. Secukinumab in PFS for s.c. self-administration Q4W.
Period: Overall Study
Arm/Group | Secukinumab (AIN457) 75mg Group 1 | Secukinumab (AIN457) 150mg Group 2 | Pbo in Core Then AIN457 75mg Group 1 | Pbo in Core Then AIN457 150mg Group 2
Started | 100 | 87 | 46 | 41
Completed | 87 | 75 | 35 | 33
Not Completed | 13 | 12 | 11 | 8
Not completed — Adverse Event | 2 | 0 | 3 | 3
Not completed — Lack of Efficacy | 1 | 0 | 2 | 1
Not completed — Lost to Follow-up | 2 | 2 | 1 | 1
Not completed — Physician Decision | 1 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Technical problems | 0 | 1 | 1 | 0
Not completed — Subject/guardian decision | 6 | 9 | 3 | 1
Not completed — Death | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab (AIN457) 75mg Group 1 | Secukinumab (AIN457) 150mg Group 2 | Pbo in Core Then AIN457 75mg Group 1 | Pbo in Core Then AIN457 150mg Group 2 | Total
Number analyzed (Participants) | 100 | 87 | 46 | 41 | 274
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (13.37) | 38.2 (11.58) | 43.0 (13.00) | 42.5 (12.13) | 41.2 (12.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 29 | 10 | 12 | 76
  Male | 75 | 58 | 36 | 29 | 198
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 7 | 1 | 1 | 12
  Asian | 19 | 15 | 8 | 8 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 61 | 48 | 30 | 28 | 167
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 17 | 17 | 7 | 4 | 45

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Spondyloarthritis International Society Criteria (ASAS) 20 Response From Week 104 to Week 260
Description: ASAS 20 response is a validated composite assessment, reflecting the proportion of treated patients who achieve within a defined time frame at least 20% improvement in score in at least 3 of a conventional set of 4 clinical domains relevant to AS and no worsening in the fourth domain. In this study, ASAS 20 is used to assess quantitatively the sustainability of clinical benefits of two dosage regimens of secukinumab over the treatment period from Week 104 to Week 260 No Statistical Analysis was performed This was the total for Group 1 Participants that up-titrated are counted only at the originally randomized treatment group.
Time Frame: Week 104 to Week 260
Population: Extension Full Analysis Set (FAS): all participants enrolled in the extension study. No Statistical Analysis was performed
Measure: Number; unit: % of responders
Arm/Group | Secukinumab (AIN457) 75mg Group 1 | Secukinumab (AIN457) 150mg Group 2 | Pbo in Core Then AIN457 75mg Group 1 | Pbo in Core Then AIN457 150mg Group 2
Number analyzed (Participants) | 100 | 87 | 46 | 41
% of responders
  Week 104: number analyzed (Participants) | 84 | 80 | 42 | 37
  Week 104 | 71.4 | 80.0 | 78.6 | 73.0
  Week 116: number analyzed (Participants) | 96 | 84 | 46 | 41
  Week 116 | 76.0 | 82.1 | 76.1 | 70.7
  Week 128: number analyzed (Participants) | 97 | 83 | 46 | 40
  Week 128 | 70.1 | 77.1 | 84.8 | 75.0
  Week 140: number analyzed (Participants) | 96 | 84 | 45 | 40
  Week 140 | 77.1 | 75.0 | 75.6 | 72.5
  Week 156: number analyzed (Participants) | 98 | 86 | 46 | 40
  Week 156 | 75.5 | 80.2 | 76.1 | 67.5
  Week 168: number analyzed (Participants) | 95 | 83 | 42 | 37
  Week 168 | 74.7 | 78.3 | 83.3 | 78.4
  Week 180: number analyzed (Participants) | 93 | 80 | 42 | 37
  Week 180 | 81.7 | 80.0 | 81.0 | 78.4
  Week 192: number analyzed (Participants) | 94 | 79 | 42 | 37
  Week 192 | 72.3 | 84.8 | 81.0 | 73.0
  Week 208: number analyzed (Participants) | 94 | 79 | 40 | 37
  Week 208 | 73.4 | 79.7 | 75.0 | 78.4
  Week 220: number analyzed (Participants) | 90 | 77 | 37 | 36
  Week 220 | 74.4 | 81.8 | 81.1 | 75.0
  Week 232: number analyzed (Participants) | 90 | 78 | 37 | 36
  Week 232 | 76.7 | 82.1 | 75.7 | 77.8
  Week 244: number analyzed (Participants) | 87 | 78 | 35 | 34
  Week 244 | 74.7 | 82.1 | 80.0 | 76.5
  Week 260: number analyzed (Participants) | 87 | 76 | 38 | 36
  Week 260 | 71.3 | 77.6 | 81.6 | 80.6

2. Secondary Outcome: Assessment of Spondyloarthritis International Society Criteria (ASAS) 40 Response From Week 104 to Week 260
Description: ASAS 40 response is a validated composite assessment, reflecting the proportion of treated patients who achieve within a defined time frame at least 40% improvement in score in at least 3 of a conventional set of 4 clinical domains relevant to AS and no worsening in the fourth domain. In this study, ASAS 40 is used to assess quantitatively the sustainability of clinical benefits of two dosage regimens of secukinumab over the treatment period from Week 104 to Week 260 No Statistical Analysis was performed This was the total for Group 1 Participants that up-titrated are counted only at the originally randomized treatment group
Time Frame: Week 104 to Week 260
Population: as for outcome 1
Measure: Number; unit: % of responders
Arm/Group | Secukinumab (AIN457) 75mg Group 1 | Secukinumab (AIN457) 150mg Group 2 | Pbo in Core Then AIN457 75mg Group 1 | Pbo in Core Then AIN457 150mg Group 2
Number analyzed (Participants) | 100 | 87 | 46 | 41
% of responders
  Week 104: number analyzed (Participants) | 84 | 80 | 42 | 37
  Week 104 | 53.6 | 65.0 | 57.1 | 48.6
  Week 116: number analyzed (Participants) | 96 | 84 | 46 | 41
  Week 116 | 56.3 | 59.5 | 54.3 | 51.2
  Week 128: number analyzed (Participants) | 97 | 83 | 46 | 40
  Week 128 | 54.6 | 68.7 | 58.7 | 55.0
  Week 140: number analyzed (Participants) | 96 | 84 | 45 | 40
  Week 140 | 53.1 | 60.7 | 53.3 | 60.0
  Week 156: number analyzed (Participants) | 98 | 86 | 46 | 40
  Week 156 | 50.0 | 62.8 | 54.3 | 55.0
  Week 168: number analyzed (Participants) | 95 | 83 | 42 | 37
  Week 168 | 54.7 | 67.5 | 42.9 | 62.2
  Week 180: number analyzed (Participants) | 93 | 80 | 42 | 37
  Week 180 | 52.7 | 68.8 | 52.4 | 67.6
  Week 192: number analyzed (Participants) | 94 | 79 | 42 | 37
  Week 192 | 57.4 | 69.6 | 52.4 | 62.2
  Week 208: number analyzed (Participants) | 94 | 79 | 40 | 37
  Week 208 | 52.1 | 60.8 | 62.5 | 56.8
  Week 220: number analyzed (Participants) | 90 | 77 | 37 | 36
  Week 220 | 51.1 | 67.5 | 54.1 | 63.9
  Week 232: number analyzed (Participants) | 90 | 78 | 37 | 36
  Week 232 | 62.2 | 66.7 | 59.5 | 69.4
  Week 244: number analyzed (Participants) | 87 | 78 | 35 | 34
  Week 244 | 60.9 | 70.5 | 62.9 | 61.8
  Week 260: number analyzed (Participants) | 87 | 76 | 38 | 36
  Week 260 | 50.6 | 64.5 | 63.2 | 66.7

ADVERSE EVENTS:
Time Frame: CAIN457F2305 (Wk 0 to Wk 104)- Cumuilative & Wk 104E1 to Wk 260 for CAIN457F2305E1
Description: Safety includes cumulative data for core & extension for patients who continued in the extension.
Groups:
- Any Secukinumab (AIN457) 75 mg: Any Secukinumab (AIN457) 75 mg safety in Core Study CAIN457F2305 and this extension study.
- Any Secukinumab (AIN457) 150 mg: Any Secukinumab (AIN457) 150 mgsafety in Core Study CAIN457F2305 and this extension study
- Placebo: Placebo in Core study CAIN457F2305E1
Arm/Group | Any Secukinumab (AIN457) 75 mg | Any Secukinumab (AIN457) 150 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 2/179 | 1/263 | 1/122
Serious Adverse Events (participants affected / at risk) | 36/179 | 33/263 | 5/122
Other Adverse Events (participants affected / at risk) | 126/179 | 157/263 | 45/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any Secukinumab (AIN457) 75 mg (N=179) | Any Secukinumab (AIN457) 150 mg (N=263) | Placebo (N=122)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 2 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Cardiorenal syndrome (Cardiac disorders) | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 3 | 3 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 1 | 1 | 0
Iridocyclitis (Eye disorders) | 0 | 2 | 0
Uveitis (Eye disorders) | 0 | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 2 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Lumbar hernia (Gastrointestinal disorders) | 1 | 0 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 1
Application site pain (General disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 3 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 2 | 0 | 0
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0
Helicobacter gastritis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0
Pulmonary tuberculoma (Infections and infestations) | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 2 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 2 | 0
Embolic stroke (Nervous system disorders) | 0 | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0
Stroke in evolution (Nervous system disorders) | 1 | 0 | 0
Trigeminal neuralgia (Nervous system disorders) | 1 | 0 | 0
Vocal cord paresis (Nervous system disorders) | 0 | 0 | 1
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Device failure (Product Issues) | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Peripheral venous disease (Vascular disorders) | 1 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any Secukinumab (AIN457) 75 mg (N=179) | Any Secukinumab (AIN457) 150 mg (N=263) | Placebo (N=122)
Leukopenia (Blood and lymphatic system disorders) | 14 | 11 | 1
Uveitis (Eye disorders) | 10 | 15 | 2
Abdominal pain upper (Gastrointestinal disorders) | 9 | 9 | 0
Diarrhoea (Gastrointestinal disorders) | 26 | 29 | 7
Mouth ulceration (Gastrointestinal disorders) | 10 | 8 | 3
Nausea (Gastrointestinal disorders) | 12 | 12 | 2
Bronchitis (Infections and infestations) | 9 | 17 | 2
Gastroenteritis (Infections and infestations) | 10 | 10 | 1
Influenza (Infections and infestations) | 19 | 26 | 2
Nasopharyngitis (Infections and infestations) | 45 | 63 | 9
Pharyngitis (Infections and infestations) | 13 | 24 | 1
Rhinitis (Infections and infestations) | 6 | 14 | 0
Upper respiratory tract infection (Infections and infestations) | 29 | 21 | 2
Urinary tract infection (Infections and infestations) | 10 | 12 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 18 | 14 | 5
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 11 | 13 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 24 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 20 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 9 | 5 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 7 | 2
Headache (Nervous system disorders) | 26 | 28 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 18 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 | 18 | 6
Hypertension (Vascular disorders) | 13 | 11 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety

DOCUMENTS (2):
  • Study Protocol (2015-08-31): https://cdn.clinicaltrials.gov/large-docs/32/NCT01863732/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/32/NCT01863732/SAP_001.pdf